CLINICAL TRIAL: NCT02920411
Title: Estudio Piloto Sobre la Efectividad de la acción Conjunta de Una Crema Corporal y un bálsamo Corporal en niños Con Dermatitis atópica
Brief Title: Effectiveness of a Combined Dermatological Treatment in Children With Atopic Dermatitis
Acronym: KAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Clever Instruments S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAOS-02-16
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined dermatological treatment (Experimental): A combined treatment of two emollient products will be applied:
  * Pediatopic treatment cream during acute stages of atopic dermatitis and
  * Pediatopic body lotion during stable stages
  Interventions: Other: Pediatopic Treatment Cream; Other: Pediatopic Body lotion

INTERVENTIONS:
Other: Pediatopic Treatment Cream — Applied twice a day minimum.
Other: Pediatopic Body lotion — Applied at libitum.

SUMMARY:
The purpose of this study is to determine the effectiveness of a combined dermatological treatment in children up to 5 years old with mild or moderated atopic dermatitis.

DETAILED DESCRIPTION:
The intensive cream and body lotion of the PediATOPIC® products are two emollients expressly formulated to serve as adjuvants in the management of Atopic Dermatitis. Both products contain Dermosense complex®, a complex that includes 3 products: Bodyfensine peptide® (inductor of dephensine synthesis against microbial aggressions), Unimoist® (the mimetizing complex of the skin's natural hydration factor), and Ramnosoft® (polysaccharide that inhibits the adhesion of pro-inflammatory drugs and bacteria, while limiting the spread of inflammatory reactions in skin cells). They also contain Bisabolol, (plant extract with anti-inflammatory, anti-irritant and antimicrobial properties) and Panthenol (Pro vitamin B5 that accelerates the skin's natural regeneration process).

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 month to 5 years old
* Patients with atopic dermatitis mild-moderate with an SCORAD=16-40

Exclusion Criteria:

* Other dermatological diseases that could interfere with the study results
* Corticoids use during 3 weeks prior to the study
* Antibiotics use to treat atopic dermatitis during 3 weeks prior to the study
* Use of topical immunomodulators
* Concurrent use of other emollients

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Changes in Atopic Dermatitis severity according SCORAD test | At 15 days
  <16 mild; >16<40 moderate; >40 severe

SECONDARY OUTCOMES:
Number of atopic dermatitis outbreaks | At 5 months
  Number of episodes
Duration of stable periods (between outbreaks) | At 5 months
  Register of days without outbreaks
Patient satisfaction assessed by Visual Analog Scales | At 5 months
  Validated scale for patients <5 years
Treatment compliance assessed by Morisky-Green test | At 5 months
  Adherence / Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Sapena Jordi, MD, Principal Investigator — Centro Médico Quirón Teknon; M.Carmen Gavilan, MD, Principal Investigator — Centro Digest Pediatric Badalona
Locations (2):
- Spain (2):
  - Centre Medic Digest, Badalona, Barcelona
  - Centro médico Quirón Teknon, Barcelona

IPD SHARING:
Plan to Share IPD: No